CLINICAL TRIAL: NCT05823012
Title: A Phase 2, Multicenter, Non-Randomized, Open-Label, Single Arm, Self-controlled Study of XP-8121 For the Treatment of Adult Subjects With Hypothyroidism
Brief Title: Study of XP-8121 For the Treatment of Adult Subjects With Hypothyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XP-8121-120
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XP-8121 (Experimental): XP-8121 100 to 1500 μg subcutaneous injection
  Interventions: Drug: levothyroxine sodium

INTERVENTIONS:
Drug: levothyroxine sodium — Levothyroxine sodium 10 mg/mL
  Other Names: XP-8121

SUMMARY:
This is a non-randomized, open-label, single arm, self-controlled study of XP-8121 (levothyroxine sodium) to determine a target dose conversion factor from stably dosed oral levothyroxine to XP-8121 (levothyroxine sodium) in patients with hypothyroidism and to assess the safety and tolerability of XP-8121(levothyroxine sodium) after once weekly subcutaneous injections. This study includes the following periods: Screening, Titration Period, and Maintenance Period. The study will conclude with an End of Maintenance Visit or Early Termination (ET) Visit.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, single arm, self-controlled study of XP-8121 (levothyroxine sodium) to determine a target dose conversion factor from stably dosed oral levothyroxine to XP-8121 (levothyroxine sodium) in patients with hypothyroidism and to assess the safety and tolerability of XP-8121 (levothyroxine sodium) after once weekly subcutaneous injections. This study includes the following periods: Screening, Titration Period (2 to 8 weeks), and Maintenance Period (4 weeks). A pharmacokinetic substudy will be conducted for a subset of participants during the Maintenance Period. The study will conclude with an End of Maintenance Visit or Early Termination (ET) Visit.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Male or female between the ages of 18 and 65 years (inclusive) at Screening, with chronic hypothyroidism and on a stable dose of oral levothyroxine (Synthroid or an FDA-approved generic equivalent to Synthroid) or, if in the pharmacokinetic substudy, Synthroid only for at least 3 months.
* Thyroid stimulating hormone (TSH) within the normal range at Screening (central laboratory) and at least 3 months prior to Screening (documented by local laboratory).
* Free thyroxine within the normal range at Screening (central laboratory).

Exclusion Criteria:

* History of hypersensitivity to levothyroxine (any formulation).
* Current dose of oral levothyroxine, based on body weight >2 μg/kg/day.
* Current levothyroxine total daily dose either <50 μg or >375 μg.
* Current use of combined thyroid treatment (i.e., Synthroid plus liothyronine or Synthroid plus Armour Thyroid) and/or any other levothyroxine aside from those used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Conoscenti, MD, Study Director — Xeris Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - ProSciento, Inc., Chula Vista, California
  - Catalina Research Institute, L.L.C., Montclair, California
  - Panax Clinical Research, LLC, Miami Lakes, Florida
  - American Research Corporation, San Antonio, Texas
  - Mt. Olympus Medical Research, LLC, Sugar Land, Texas
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited over an approximate 7.5 month period at medical research centers with experience in hypothyroidism.
Pre-assignment Details: A total of 140 potential participants were screened, 46 participants were enrolled, and 94 potential participants were screen failures. The most common reasons for screen failure were fT4 and TSH outside of the normal range as required by the eligibility criteria.
Groups:
- XP-8121: All participants who received at least 1 dose of XP-8121 (100 to 1500 μg subcutaneous injection).
Period: Titration Period
Arm/Group | XP-8121
Started | 46
Completed | 42
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Inability to Achieve a tolerable replacement dosage | 3
Period: Maintenance Period
Arm/Group | XP-8121
Started | 42
Completed | 39
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Inability to achieve a tolerable replacement dosage | 1
Not completed — Inability to achieve an adequate replacement dosage | 1

BASELINE CHARACTERISTICS:
Arm/Group | XP-8121
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 54.5 [33 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 1
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Baseline Body Mass Index [Median (Full Range); unit: kg/m^2] — Screening eligibility criteria required a BMI of 18 to 40 kg/m^2.
  kg/m^2 | 29.50 [23.1 to 39.9]
Primary Hypothyroidism History [Count of Participants; unit: Participants] | 46
Prior Daily Oral Levothyroxine Brand [Count of Participants; unit: Participants]
  Synthroid | 9
  Other Brand or Generic | 37
Prior Daily Oral Levothyroxine Dose [Count of Participants; unit: Participants]
  50 micrograms | 14
  75 micrograms | 12
  88 micrograms | 3
  100 micrograms | 8
  112 micrograms | 3
  125 micrograms | 3
  150 micrograms | 2
  175 micrograms | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose Conversion Factor
Description: Geometric mean ratio of the weekly dose of XP-8121 to the daily dose of oral levothyroxine (aka dose conversion factor), where the XP-8121 dose corresponds to the administration immediately preceding collection of blood TSH used to determine normalization at the end of Maintenance Period. The dose conversion factor was assessed by comparing the natural log-transformed final XP-8121 dose in μg that maintained normalized TSH throughout the Maintenance Period to the natural log-transformed daily oral levothyroxine dose the participant was taking before the study, using a linear mixed effects model with treatment as the fixed effect and subject as the random effect. Geometric least square means (LSMs) were calculated by exponentiating the LSM from the ANOVA. The geometric mean ratio and the corresponding 90% CI was found by exponentiating the differences of log-transformed LSM and 90% confidence interval (CI) of the difference.
Time Frame: Day 29 of the Maintenance Period
Population: The Completer Population used for this analysis is defined as all participants who completed the Maintenance Period and exhibited normalized TSH throughout the Maintenance Period while on a stable dose of XP-8121 for approximately 6 weeks. Participants with a reduced dose at any point during the Maintenance Period were not included in the Completer Population.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | XP-8121
Number analyzed (Participants) | 23
Ratio | 4.24 [4.06 to 4.42]

2. Primary Outcome: Tolerability Assessment: Modified Draize Scale - Erythema
Description: The Modified Draize Scale assessment of erythema and edema was conducted 30 (+/-5) minutes after each dosing. The Modified Draize Scale is a 5-point scale: 0-none, 1-very slight, 2-slight, 3-moderate, 4-severe.
Time Frame: Week 1 Dosing in Titration Period through Day 22 Dosing in Maintenance Period
Population: The number of participants at each timepoint is dependent on the number of participants dosed at each timepoint. The number of participants decreases in association with study withdrawal, with the exception of the reduction in the number of participants in Titration Periods Week 7 and Week 8 due to the number of participants that transitioned to the Maintenance Period after dosing at Week 6.
Measure: Count of Participants; unit: Participants
Arm/Group | XP-8121
Number analyzed (Participants) | 46
Participants
  Titration Period: Week 1 Dosing: 0 - None | 43
  Titration Period: Week 1 Dosing: 1 - Very Slight | 3
  Titration Period: Week 1 Dosing: 2 - Slight | 0
  Titration Period: Week 1 Dosing: 3 - Moderate | 0
  Titration Period: Week 1 Dosing: 4 - Severe | 0
  Titration Period: Week 2 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 2 Dosing: 0 - None | 41
  Titration Period: Week 2 Dosing: 1 - Very Slight | 2
  Titration Period: Week 2 Dosing: 2 - Slight | 0
  Titration Period: Week 2 Dosing: 3 - Moderate | 0
  Titration Period: Week 2 Dosing: 4 - Severe | 0
  Titration Period: Week 3 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 3 Dosing: 0 - None | 41
  Titration Period: Week 3 Dosing: 1 - Very Slight | 2
  Titration Period: Week 3 Dosing: 2 - Slight | 0
  Titration Period: Week 3 Dosing: 3 - Moderate | 0
  Titration Period: Week 3 Dosing: 4 - Severe | 0
  Titration Period: Week 4 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 4 Dosing: 0 - None | 37
  Titration Period: Week 4 Dosing: 1 - Very Slight | 5
  Titration Period: Week 4 Dosing: 2 - Slight | 0
  Titration Period: Week 4 Dosing: 3 - Moderate | 0
  Titration Period: Week 4 Dosing: 4 - Severe | 0
  Titration Period: Week 5 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 5 Dosing: 0 - None | 38
  Titration Period: Week 5 Dosing: 1 - Very Slight | 4
  Titration Period: Week 5 Dosing: 2 - Slight | 0
  Titration Period: Week 5 Dosing: 3 - Moderate | 0
  Titration Period: Week 5 Dosing: 4 - Severe | 0
  Titration Period: Week 6 Dosing: number analyzed (Participants) | 41
  Titration Period: Week 6 Dosing: 0 - None | 38
  Titration Period: Week 6 Dosing: 1 - Very Slight | 3
  Titration Period: Week 6 Dosing: 2 - Slight | 0
  Titration Period: Week 6 Dosing: 3 - Moderate | 0
  Titration Period: Week 6 Dosing: 4 - Severe | 0
  Titration Period: Week 7 Dosing: number analyzed (Participants) | 13
  Titration Period: Week 7 Dosing: 0 - None | 12
  Titration Period: Week 7 Dosing: 1 - Very Slight | 1
  Titration Period: Week 7 Dosing: 2 - Slight | 0
  Titration Period: Week 7 Dosing: 3 - Moderate | 0
  Titration Period: Week 7 Dosing: 4 - Severe | 0
  Titration Period: Week 8 Dosing: number analyzed (Participants) | 12
  Titration Period: Week 8 Dosing: 0 - None | 12
  Titration Period: Week 8 Dosing: 1 - Very Slight | 0
  Titration Period: Week 8 Dosing: 2 - Slight | 0
  Titration Period: Week 8 Dosing: 3 - Moderate | 0
  Titration Period: Week 8 Dosing: 4 - Severe | 0
  Maintenance Period: Day 1 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 1 Dosing: 0 - None | 40
  Maintenance Period: Day 1 Dosing: 1 - Very Slight | 2
  Maintenance Period: Day 1 Dosing: 2 - Slight | 0
  Maintenance Period: Day 1 Dosing: 3 - Moderate | 0
  Maintenance Period: Day 1 Dosing: 4 - Severe | 0
  Maintenance Period: Day 8 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 8 Dosing: 0 - None | 40
  Maintenance Period: Day 8 Dosing: 1 - Very Slight | 2
  Maintenance Period: Day 8 Dosing: 2 - Slight | 0
  Maintenance Period: Day 8 Dosing: 3 - Moderate | 0
  Maintenance Period: Day 8 Dosing: 4 - Severe | 0
  Maintenance Period: Day 15 Dosing: number analyzed (Participants) | 41
  Maintenance Period: Day 15 Dosing: 0 - None | 39
  Maintenance Period: Day 15 Dosing: 1 - Very Slight | 1
  Maintenance Period: Day 15 Dosing: 2 - Slight | 1
  Maintenance Period: Day 15 Dosing: 3 - Moderate | 0
  Maintenance Period: Day 15 Dosing: 4 - Severe | 0
  Maintenance Period: Day 22 Dosing: number analyzed (Participants) | 39
  Maintenance Period: Day 22 Dosing: 0 - None | 37
  Maintenance Period: Day 22 Dosing: 1 - Very Slight | 2
  Maintenance Period: Day 22 Dosing: 2 - Slight | 0
  Maintenance Period: Day 22 Dosing: 3 - Moderate | 0
  Maintenance Period: Day 22 Dosing: 4 - Severe | 0

3. Primary Outcome: Tolerability Assessment: Modified Draize Scale - Edema
Description: as for outcome 2
Time Frame: Week 1 Dosing in Titration Period through Day 22 Dosing in Maintenance Period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | XP-8121
Number analyzed (Participants) | 46
Participants
  Titration Period: Week 1 Dosing: 0 - None | 44
  Titration Period: Week 1 Dosing: 1 - Very Slight | 2
  Titration Period: Week 1 Dosing: 2 - Slight | 0
  Titration Period: Week 1 Dosing: 3 - Moderate | 0
  Titration Period: Week 1 Dosing: 4 - Severe | 0
  Titration Period: Week 2 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 2 Dosing: 0 - None | 43
  Titration Period: Week 2 Dosing: 1 - Very Slight | 0
  Titration Period: Week 2 Dosing: 2 - Slight | 0
  Titration Period: Week 2 Dosing: 3 - Moderate | 0
  Titration Period: Week 2 Dosing: 4 - Severe | 0
  Titration Period: Week 3 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 3 Dosing: 0 - None | 43
  Titration Period: Week 3 Dosing: 1 - Very Slight | 0
  Titration Period: Week 3 Dosing: 2 - Slight | 0
  Titration Period: Week 3 Dosing: 3 - Moderate | 0
  Titration Period: Week 3 Dosing: 4 - Severe | 0
  Titration Period: Week 4 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 4 Dosing: 0 - None | 41
  Titration Period: Week 4 Dosing: 1 - Very Slight | 1
  Titration Period: Week 4 Dosing: 2 - Slight | 0
  Titration Period: Week 4 Dosing: 3 - Moderate | 0
  Titration Period: Week 4 Dosing: 4 - Severe | 0
  Titration Period: Week 5 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 5 Dosing: 0 - None | 42
  Titration Period: Week 5 Dosing: 1 - Very Slight | 0
  Titration Period: Week 5 Dosing: 2 - Slight | 0
  Titration Period: Week 5 Dosing: 3 - Moderate | 0
  Titration Period: Week 5 Dosing: 4 - Severe | 0
  Titration Period: Week 6 Dosing: number analyzed (Participants) | 41
  Titration Period: Week 6 Dosing: 0 - None | 41
  Titration Period: Week 6 Dosing: 1 - Very Slight | 0
  Titration Period: Week 6 Dosing: 2 - Slight | 0
  Titration Period: Week 6 Dosing: 3 - Moderate | 0
  Titration Period: Week 6 Dosing: 4 - Severe | 0
  Titration Period: Week 7 Dosing: number analyzed (Participants) | 13
  Titration Period: Week 7 Dosing: 0 - None | 11
  Titration Period: Week 7 Dosing: 1 - Very Slight | 1
  Titration Period: Week 7 Dosing: 2 - Slight | 1
  Titration Period: Week 7 Dosing: 3 - Moderate | 0
  Titration Period: Week 7 Dosing: 4 - Severe | 0
  Titration Period: Week 8 Dosing: number analyzed (Participants) | 12
  Titration Period: Week 8 Dosing: 0 - None | 12
  Titration Period: Week 8 Dosing: 1 - Very Slight | 0
  Titration Period: Week 8 Dosing: 2 - Slight | 0
  Titration Period: Week 8 Dosing: 3 - Moderate | 0
  Titration Period: Week 8 Dosing: 4 - Severe | 0
  Maintenance Period: Day 1 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 1 Dosing: 0 - None | 42
  Maintenance Period: Day 1 Dosing: 1 - Very Slight | 0
  Maintenance Period: Day 1 Dosing: 2 - Slight | 0
  Maintenance Period: Day 1 Dosing: 3 - Moderate | 0
  Maintenance Period: Day 1 Dosing: 4 - Severe | 0
  Maintenance Period: Day 8 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 8 Dosing: 0 - None | 42
  Maintenance Period: Day 8 Dosing: 1 - Very Slight | 0
  Maintenance Period: Day 8 Dosing: 2 - Slight | 0
  Maintenance Period: Day 8 Dosing: 3 - Moderate | 0
  Maintenance Period: Day 8 Dosing: 4 - Severe | 0
  Maintenance Period: Day 15 Dosing: number analyzed (Participants) | 41
  Maintenance Period: Day 15 Dosing: 0 - None | 40
  Maintenance Period: Day 15 Dosing: 1 - Very Slight | 0
  Maintenance Period: Day 15 Dosing: 2 - Slight | 1
  Maintenance Period: Day 15 Dosing: 3 - Moderate | 0
  Maintenance Period: Day 15 Dosing: 4 - Severe | 0
  Maintenance Period: Day 22 Dosing: number analyzed (Participants) | 39
  Maintenance Period: Day 22 Dosing: 0 - None | 39
  Maintenance Period: Day 22 Dosing: 1 - Very Slight | 0
  Maintenance Period: Day 22 Dosing: 2 - Slight | 0
  Maintenance Period: Day 22 Dosing: 3 - Moderate | 0
  Maintenance Period: Day 22 Dosing: 4 - Severe | 0

4. Primary Outcome: Tolerability Assessments: Injection Site Discomfort Evaluation
Description: Injection site discomfort was assessed by each participant at 10 (+/-2) minutes post-injection.
Time Frame: Week 1 dosing in the Titration Period through Day 22 dosing in the Maintenance Period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | XP-8121
Number analyzed (Participants) | 46
Participants
  Titration Period: Week 1 Dosing: Yes | 14
  Titration Period: Week 1 Dosing: No | 32
  Titration Period: Week 2 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 2 Dosing: Yes | 9
  Titration Period: Week 2 Dosing: No | 34
  Titration Period: Week 3 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 3 Dosing: Yes | 12
  Titration Period: Week 3 Dosing: No | 31
  Titration Period: Week 4 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 4 Dosing: Yes | 10
  Titration Period: Week 4 Dosing: No | 32
  Titration Period: Week 5 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 5 Dosing: Yes | 12
  Titration Period: Week 5 Dosing: No | 30
  Titration Period: Week 6 Dosing: number analyzed (Participants) | 41
  Titration Period: Week 6 Dosing: Yes | 9
  Titration Period: Week 6 Dosing: No | 32
  Titration Period: Week 7 Dosing: number analyzed (Participants) | 13
  Titration Period: Week 7 Dosing: Yes | 6
  Titration Period: Week 7 Dosing: No | 7
  Titration Period: Week 8 Dosing: number analyzed (Participants) | 12
  Titration Period: Week 8 Dosing: Yes | 2
  Titration Period: Week 8 Dosing: No | 10
  Maintenance Period: Day 1 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 1 Dosing: Yes | 13
  Maintenance Period: Day 1 Dosing: No | 29
  Maintenance Period: Day 8 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 8 Dosing: Yes | 12
  Maintenance Period: Day 8 Dosing: No | 30
  Maintenance Period: Day 15 Dosing: number analyzed (Participants) | 41
  Maintenance Period: Day 15 Dosing: Yes | 8
  Maintenance Period: Day 15 Dosing: No | 33
  Maintenance Period: Day 22 Dosing: number analyzed (Participants) | 39
  Maintenance Period: Day 22 Dosing: Yes | 6
  Maintenance Period: Day 22 Dosing: No | 33

5. Secondary Outcome: Proportion of Participants With Normalized TSH Throughout the Maintenance Period
Description: Proportion of participants enrolled with normalized TSH throughout the Maintenance Period
Time Frame: Day 29 of the Maintenance Period
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants who received at least 1 dose of XP-8121 (100 to 1500 μg subcutaneous injection).
- Participants Who Entered the Maintenance Period: All participants who received XP-8121 (100 to 1500 μg subcutaneous injection), completed the Titration Period, and entered the Maintenance Period.
Arm/Group | All Participants | Participants Who Entered the Maintenance Period
Number analyzed (Participants) | 46 | 42
Participants | 27 | 27

6. Secondary Outcome: Proportion of Participants With Normalized TSH at End of Maintenance Period
Description: Proportion of participants enrolled with normalized TSH at the end of the Maintenance Period.
Time Frame: Day 29 of the Maintenance Period
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Entered Maintenance Period: All participants who received XP-8121 (100 to 1500 μg subcutaneous injection), completed the Titration Period, and entered the Maintenance Period.
Arm/Group | All Participants | Participants Who Entered Maintenance Period
Number analyzed (Participants) | 46 | 42
Participants | 31 | 31

7. Secondary Outcome: Thyroid Hormone Concentrations: Total Thyroxine
Description: Thyroid hormone concentrations (total thyroxine, free protein-unbound thyroxine (fT4), and TSH) following the first dose of XP-8121 during the Titration Period and Maintenance Periods
Time Frame: Up to Day 29 of the Maintenance Period
Population: The number of participants at each timepoint is dependent on the number of participants dosed at each timepoint. The overall number follows the decrease associated with study withdrawal, with the exception of the reduction in the number of participants in Titration Periods Week 7 and Week 8 due to the number of participants that transitioned to the Maintenance Period after dosing at Week 6.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | XP-8121
Number analyzed (Participants) | 46
nmol/L
  Titration Period: Baseline | 103.68 (27.278)
  Titration Period: Week 2 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 2 Dosing | 88.17 (23.019)
  Titration Period: Week 3 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 3 Dosing | 89.68 (23.019)
  Titration Period: Week 4 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 4 Dosing | 92.44 (24.104)
  Titration Period: Week 5 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 5 Dosing | 94.26 (22.059)
  Titration Period: Week 6 Dosing: number analyzed (Participants) | 39
  Titration Period: Week 6 Dosing | 97.38 (22.056)
  Titration Period: Week 7 Dosing: number analyzed (Participants) | 13
  Titration Period: Week 7 Dosing | 90.29 (18.867)
  Titration Period: Week 8 Dosing: number analyzed (Participants) | 12
  Titration Period: Week 8 Dosing | 88.58 (25.032)
  Maintenance Period: Day 1 Dosing (Baseline): number analyzed (Participants) | 42
  Maintenance Period: Day 1 Dosing (Baseline) | 103.45 (24.970)
  Maintenance Period: Day 8 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 8 Dosing | 102.24 (23.704)
  Maintenance Period: Day 15 Dosing: number analyzed (Participants) | 41
  Maintenance Period: Day 15 Dosing | 103.35 (23.508)
  Maintenance Period: Day 22 Dosing: number analyzed (Participants) | 38
  Maintenance Period: Day 22 Dosing | 104.67 (19.389)
  Maintenance Period: Day 29: number analyzed (Participants) | 39
  Maintenance Period: Day 29 | 101.97 (24.532)

8. Secondary Outcome: Thyroid Hormone Concentrations: Free Thyroxine (fT4)
Description: as for outcome 7
Time Frame: Up to Day 29 of the Maintenance Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | XP-8121
Number analyzed (Participants) | 46
pmol/L
  Titration Period: Baseline | 14.60 (2.713)
  Titration Period: Week 2 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 2 Dosing | 12.09 (2.209)
  Titration Period: Week 3 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 3 Dosing | 11.69 (2.494)
  Titration Period: Week 4 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 4 Dosing | 12.47 (2.668)
  Titration Period: Week 5 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 5 Dosing | 12.84 (2.417)
  Titration Period: Week 6 Dosing: number analyzed (Participants) | 39
  Titration Period: Week 6 Dosing | 12.88 (1.977)
  Titration Period: Week 7 Dosing: number analyzed (Participants) | 13
  Titration Period: Week 7 Dosing | 12.32 (1.814)
  Titration Period: Week 8 Dosing: number analyzed (Participants) | 12
  Titration Period: Week 8 Dosing | 13.26 (1.840)
  Maintenance Period: Day 1 Dosing (Baseline): number analyzed (Participants) | 42
  Maintenance Period: Day 1 Dosing (Baseline) | 14.50 (2.411)
  Maintenance Period: Day 8 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 8 Dosing | 14.36 (2.319)
  Maintenance Period: Day 15 Dosing: number analyzed (Participants) | 41
  Maintenance Period: Day 15 Dosing | 14.24 (2.147)
  Maintenance Period: Day 22 Dosing: number analyzed (Participants) | 38
  Maintenance Period: Day 22 Dosing | 14.27 (1.917)
  Maintenance Period: Day 29: number analyzed (Participants) | 39
  Maintenance Period: Day 29 | 14.14 (1.796)

9. Secondary Outcome: Thyroid Hormone Concentrations: Thyroid Stimulating Hormone (TSH)
Description: as for outcome 7
Time Frame: Up to Day 29 of the Maintenance Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | XP-8121
Number analyzed (Participants) | 46
mIU/L
  Titration Period: Baseline | 1.958 (1.0778)
  Titration Period: Week 2 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 2 Dosing | 3.942 (2.8299)
  Titration Period: Week 3 Dosing: number analyzed (Participants) | 43
  Titration Period: Week 3 Dosing | 6.534 (8.2589)
  Titration Period: Week 4 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 4 Dosing | 6.162 (8.8632)
  Titration Period: Week 5 Dosing: number analyzed (Participants) | 42
  Titration Period: Week 5 Dosing | 6.397 (9.8016)
  Titration Period: Week 6 Dosing: number analyzed (Participants) | 39
  Titration Period: Week 6 Dosing | 5.506 (7.1427)
  Titration Period: Week 7 Dosing: number analyzed (Participants) | 13
  Titration Period: Week 7 Dosing | 8.326 (8.5120)
  Titration Period: Week 8 Dosing: number analyzed (Participants) | 12
  Titration Period: Week 8 Dosing | 5.752 (5.3967)
  Maintenance Period: Day 1 Dosing (Baseline): number analyzed (Participants) | 42
  Maintenance Period: Day 1 Dosing (Baseline) | 2.967 (2.1827)
  Maintenance Period: Day 8 Dosing: number analyzed (Participants) | 42
  Maintenance Period: Day 8 Dosing | 2.920 (2.7009)
  Maintenance Period: Day 15 Dosing: number analyzed (Participants) | 41
  Maintenance Period: Day 15 Dosing | 2.739 (2.8858)
  Maintenance Period: Day 22 Dosing: number analyzed (Participants) | 38
  Maintenance Period: Day 22 Dosing | 2.494 (2.0766)
  Maintenance Period: Day 29: number analyzed (Participants) | 39
  Maintenance Period: Day 29 | 2.493 (1.5087)

ADVERSE EVENTS:
Time Frame: From Screening through the End of Maintenance Visit (Day 29) or up to 14 (+/-2 days) after last dose of XP-8121 for participants who withdrew prematurely
Groups:
- Titration Period: All participants who received at least 1 dose of XP-8121 (100 to 1500 μg subcutaneous injection) during the Titration Period.
- Maintenance Period: All participants who received at least 1 dose of XP-8121 (100 to 1500 μg subcutaneous injection) during the Maintenance Period. Includes only includes those participants that completed the Titration Period and entered the Maintenance Period.
- Overall: Includes all participants that received XP-8121 (100 to 1500 μg subcutaneous injection) in both Titration and Maintenance Treatment Periods.
Arm/Group | Titration Period | Maintenance Period | Overall
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/42 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/42 | 0/46
Other Adverse Events (participants affected / at risk) | 19/46 | 4/42 | 22/46
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titration Period (N=46) | Maintenance Period (N=42) | Overall (N=46)
Fatigue (General disorders) | 10 (12) | 0 (0) | 10 (12)
Injection site pain (General disorders) | 3 (4) | 2 (2) | 5 (6)
Temperature intolerance (General disorders) | 2 (3) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Weight increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 0 (0) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (5) | 1 (1) | 2 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication policy allows the Sponsor to submit a multi-center publication within 18-month period after the study is completed at all institutions. If it is not submitted within such 18-month period, an individual PI may furnish the Sponsor with a copy of any proposed publication or release at least 90 days in advance of the proposed submission or presentation. The Sponsor may review such proposed publication or release and may request a delay in publication of up to an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2023-05-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT05823012/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT05823012/SAP_001.pdf